CLINICAL TRIAL: NCT00691366
Title: Autonomic Nervous System Physiology and Chronic Pruritus: A Comprehensive Investigation of Heart Rate Variability as a Measure of the Autonomic Nervous System in Atopic Dermatitis
Brief Title: Comprehensive Investigation of Heart Rate Variability as a Measure of the Autonomic Nervous System in Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: 00002115
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2008-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to study heart rate patterns in people with moderate to severe atopic dermatitis and how itching affects those patterns.

DETAILED DESCRIPTION:
To comprehensively evaluate the autonomic nervous system through heart rate variability (HRV) measurements in patients with moderate to severe atopic dermatitis suffering from pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women who are between 18 and 50 years of age.
* Diagnosis of moderate to severe atopic dermatitis confirmed by published consensus diagnostic criteria26 (except for healthy control subjects). Severity will be based on an investigator's global assessment score and will have to be moderate or severe (IGA) (see Appendix 1).
* Subjects must be in general good health with no other skin disease, disease state or physical condition which would impair evaluation of their skin or which would increase their health risk by study participation as determined by the investigators.
* Women of child bearing potential will be required to have a negative pregnancy test in order to enroll in the study and will be required to maintain adequate birth control throughout the study. Reliable methods of birth control are: abstinence, oral contraceptives, intrauterine device (IUD), DepoProvera, Norplant, tubal ligation, or vasectomy of the partner (with confirmed negative sperm counts) in a monogamous relationship. An acceptable, although less reliable, method involves the careful use of condoms and spermicidal foam or gel and/or a cervical cap or sponge.
* Subjects must cease using topical agents on the forearm where experimental data is going to be collected at least 1 week prior. Topical agents can be used on all other parts of the body.
* Subjects will be required to cease use of oral antihistamines for a period of one week prior to and during the study visit.

Exclusion Criteria:

* Adults over age 50.
* Children less than 18 years of age.
* Unable to complete the required measures.
* Diagnosis with other diseases that would affect the measurement of heart rate variability as determined by the investigators such as cardiovascular disease, hypertension, bradycardia (<60 beats per minute) and tachycardia (>100 beats per minute) amongst others.
* Diagnosis with other skin diseases that would affect the measurement of transepidermal water loss (TEWL) and skin hydration as determined by the investigators.
* Currently enrolled in any investigational study in which the subject is receiving any type of drug, biologic, or non-drug therapy and subjects undergoing treatment with another investigational drug or approved therapy for investigational use within 28 days prior to study participation.
* Consistent consumption of more than 4 caffeinated beverages per day.
* Current treatment with oral lipophilic beta blockers, antihistamines, opioids, glucocorticoids, theophylline, anticholinergic medication or inhaled beta-agonists or anticholinergics or other medications known to interfere autonomic nervous system physiology.
* Asthma/Chronic Obstructive Airways Disease or other respiratory disease.
* Neuropathy causing diseases such as uremia.
* Uncontrolled thyroid disease.
* Diabetes mellitus.
* Use of illicit drugs.
* Current diagnosis of a psychiatric disorder27;28.
* History of chronic urticaria.
* History of anaphylactic shock.
* Allergy to histamine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Wake Forest University Health Sciences Dermatology Clinic population and from appropriate IRB-approved advertising in the community.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gil Yosipovitch, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Facility: Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States